CLINICAL TRIAL: NCT06748677
Title: Prospective Cohort Study of Minimally Invasive Surgery Versus Traditional Open Surgery for Nipple Areola Preserving Mastectomy Combined with Immediate Prosthesis Reconstruction
Brief Title: Endoscopic and Robotic NSM with Immediate Prosthesis Breast Reconstruction
Acronym: EnRoNSM
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Other Study IDs: PKUPH2024Z217
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Nipple-sparing Mastectomy; Immediate Prosthesis Reconstruction; Endoscopic Surgery; Robotic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- endoscopic and robotic surgery: nipple-sparing mastectomy under endoscopic/robotic surgery combined with immediate prosthesis reconstruction
- conventional surgery: conventional nipple-sparing mastectomy combined with immediate prosthesis reconstruction

SUMMARY:
Breast cancer is the most common malignant tumor in women. Surgical treatment is the most important treatment for early breast cancer. Breast cancer resection is considered to be a destructive operation. Patients need to accept the double blow of physical and psychological loss of breast shape. Although with the change of the concept of early diagnosis and treatment of breast cancer, the breast conserving rate of breast cancer is gradually increasing in China, more than half of the patients are still unable to retain breast due to their condition. For these patients, breast reconstruction surgery is an important means to improve the postoperative breast shape. With the improvement of surgical technology, endoscopic/robotic NSM combined with immediate prosthesis breast reconstruction has been gradually developed. According to previous literature reports, it has good tumor safety and aesthetics, but it is still lack of large-scale prospective results.

This project plans to adopt a prospective cohort design, based on the large sample breast disease cohort database established by the breast center of Peking University People's Hospital, and prospectively include patients who receive NSM combined with immediate prosthesis reconstruction under endoscopy/robot and conventional surgery from January 1, 2025 to December 31, 2028. The perioperative complications, tumor safety and patient reported outcomes of the two methods were compared.

ELIGIBILITY:
Inclusion Criteria:

1. Underwent surgical treatment at Peking University People's Hospital, with hospitalization records;
2. Preoperative core needle biopsy confirmed breast cancer;
3. The clinical stage of the tumor is stage 0-IIIB; 4）cT≤5cm， cN0/cN1，M0， And there is no tumor invasion of the nipple areola complex, skin, and chest wall;

5) Intraoperative plan to use non biological patches (such as TiLoop) to partially or completely wrap the prosthesis 6) Signed agreement to participate in this study; 7) Can cooperate to complete the Patient Reported Outcome Measures (PROMs) questionnaire.

Exclusion Criteria:

1. Lack of clinical pathological data (such as imaging data, pathological data);
2. Pregnancy or lactation period;
3. Patients with metastatic breast cancer or bilateral breast cancer;
4. Have undergone breast conserving surgery/chest radiation therapy before;
5. Patients with nipple areola invasion and subsequent removal of nipple areola complex;
6. Failed to undergo curative surgery;

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective inclusion of patients who underwent minimally invasive surgery (endoscopic and robotic surgey) and conventional surgery at Peking University People's Hospital from January 1, 2025.01 to December 31, 2028.12 to preserve the NSM with immediate prosthesis breast reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 484 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative complications | 3 months
  Delayed wound healing, nipple and areola ischemia/necrosis, skin ischemia/necrosis, serum swelling, wound dehiscence/prosthesis exposure, infection, and prosthesis removal occurred within 3 months after surgery.

SECONDARY OUTCOMES:
Patient-reported Outcome Measures | 1 year
  BREAST-Q scores, higher scores mean a better outcome
local-regional recurrence | 5 years
  From research enrollment to ipsilateral breast skin, subcutaneous, chest wall, axillary, internal mammary, and supraclavicular lymph node recurrence;
Distant metastasis free survival | 5 years
  the time from enrollment in the study to the occurrence of distant recurrence and metastasis;
Disease free survival | 5 years
  the time from study enrollment to the first occurrence of the following events defined as failure, including ipsilateral local recurrence, contralateral breast cancer, distant recurrence or death from any cause.

OTHER OUTCOMES:
tumour saftey | 1 week
  Pathology of residual cavity lavage fluid; Pathology of peripheral edge tissue in breast specimens. If we can see tumour cell in the lavage fluid or breast tissue on the peripheral edge means not safety.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China